CLINICAL TRIAL: NCT03409796
Title: Assessment of Immune Activation and Tolerance in Celiac Disease During Gluten Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TIMP-GLIA-5001; U1111-1202-6708 (Other: WHO)
Record Dates: First submitted 2017-12-31; First posted 2018-01-24 (Actual); Results first posted 2020-08-18 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Celiac Disease
Keywords: Gluten Challenge
MeSH Terms: conditions — Celiac Disease | interventions — Glutens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Gluten 3 gm (Other): Gluten 3 gram (gm), powder, orally, once daily up to 14 days.
  Interventions: Dietary Supplement: Gluten
- Group B: Gluten 10 gm (Other): Gluten 10 gm, powder, orally, once daily up to 14 days.
  Interventions: Dietary Supplement: Gluten

INTERVENTIONS:
Dietary Supplement: Gluten — Gluten powder.

SUMMARY:
The primary purpose of this study is to characterize changes in gluten-specific T cells and pathology in the small intestine with specific focus on biomarkers likely to change with therapeutic celiac disease (CeD) treatment.

DETAILED DESCRIPTION:
Gluten challenge studies are used to test the effectiveness of therapies designed to prevent immune response to gluten in participants with CeD. The study will enroll approximately 20 participants. Participants will be randomly assigned (by chance, like flipping a coin) in a 1:1 ratio to one of the two treatment groups:

* Group A: Gluten 3 gm
* Group B: Gluten 10 gm

All participants will be asked to take an oral dose of gluten at the same time on Days 1 to 14 throughout the study. This multi-center trial will be conducted in the United States. The overall time to participate in this study is 10 weeks. Participants will visit to the clinic on Day -45 and will be contacted for follow-up assessment on Days 15 to 42.

ELIGIBILITY:
Inclusion Criteria:

1. Be a non-smoker who has not used tobacco- or nicotine-containing products (example, nicotine patch) for at least 6 months before Day 1 gluten administration.
2. Have well-controlled biopsy-proven CeD, compliant with a gluten-free diet (GFD) for greater than or equal to (>=) 6 months preceding screening, with resolution of CeD symptoms, normalization of CeD serology, and in the judgment of the investigator, have inactive or minimally-active disease.
3. Be HLA-DQ2.5 and/or HLA-DQ8 positive, assessed at screening. If participants have already been genotyped, results from previous testing may be used in lieu of genotyping at screening.
4. Be willing to delay a planned procedure involving the use of powerful electromagnetic fields (example, magnetic resonance imaging), until the PillCam SB 3 capsule is excreted.
5. Not undergo VCE or optical coherence tomography (OCT) if has an implanted electromedical device or a swallowing disorder.
6. Not undergo OCT if has a contraindication to the device or procedure as per reference information.

Exclusion Criteria:

1. Had major surgery and/or donated or lost 1 unit of blood (approximately 500 milliliter [mL]) within 8 weeks before the first dose of gluten.
2. Are unable to refrain from or anticipate the use of any unapproved medication, including prescription drugs, nonprescription drugs, and herbal remedies, beginning approximately 7 days before administration of the initial dose of gluten and continuing throughout the trial until the follow-up visit.
3. Consume excessive amounts of coffee, tea, cola, energy drinks, or other caffeinated beverages per day. An excessive amount is defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine).
4. Have positive IgA anti-tissue transglutaminase (tTG), IgA anti-deamidated gliadin peptide (DGP), and IgG DGP serologies at Screening.
5. Have inflammatory gastrointestinal disorders or autoimmune diseases other than CeD or autoimmune thyroid disease.
6. Have known or suspected gastrointestinal obstructions, strictures, or fistulas based on the clinical picture or pre-procedure testing and profile of the PillCam SB 3 capsule.
7. Endoscopy and intestinal biopsy are contraindicated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Johansen A, Sandve GKF, Maxwell JR, Smithson G, Sollid LM, Stamnaes J. Biopsy Proteome Score Performs Well as an Effect Measure in a Gluten Challenge Trial of Celiac Disease. Clin Gastroenterol Hepatol. 2025 Apr;23(5):758-765.e8. doi: 10.1016/j.cgh.2024.08.005. Epub 2024 Aug 30. PMID 39209203
- [Derived] Leonard MM, Silvester JA, Leffler D, Fasano A, Kelly CP, Lewis SK, Goldsmith JD, Greenblatt E, Kwok WW, McAuliffe WJ, Galinsky K, Siegelman J, Chow IT, Wagner JA, Sapone A, Smithson G. Evaluating Responses to Gluten Challenge: A Randomized, Double-Blind, 2-Dose Gluten Challenge Trial. Gastroenterology. 2021 Feb;160(3):720-733.e8. doi: 10.1053/j.gastro.2020.10.040. Epub 2020 Oct 29. PMID 33130104
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b60374db2bf003ab4a134?idFilter=%5B%22TIMP-GLIA-5001%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the Unites Stated from 24 April 2018 to 02 May 2019.
Pre-assignment Details: Participants diagnosed with celiac disease (CeD) were enrolled in a 1:1 ratio in one of the two treatment groups: 3 gram gluten per day or 10 gram gluten per day.
Groups:
- Group A: Gluten 3 Gram: Gluten 3 gram, powder, orally, once daily up to 14 days.
- Group B: Gluten 10 Gram: Gluten 10 gram, powder, orally, once daily up to 14 days.
Period: Overall Study
Arm/Group | Group A: Gluten 3 Gram | Group B: Gluten 10 Gram
Started | 9 | 7
Completed | 7 | 6
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety set consisted of all participants who were enrolled and received at least 1 dose of gluten.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Gluten 3 Gram | Group B: Gluten 10 Gram | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (18.12) | 46.0 (18.86) | 45.0 (17.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 7 | 16
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 165.12 (9.648) | 169.76 (8.074) | 167.15 (9.020)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 75.23 (17.183) | 81.36 (8.121) | 77.91 (13.918)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Small Intestine Histology Based on Villous Height to Crypt Depth (Vh:Cd) Ratio
Description: Attenuation of the effects of gluten exposure was assessed by measuring the change from baseline in villous height (Vh) to crypt depth (Cd) ratio after 15 days of gluten challenge. Villi were the small finger like projections that line the small intestine and promote nutrient absorption and are often shortened in participants with CeD. Crypts were grooves between the villi that are often elongated in participants with CeD. A decreased Vh:Cd ratio indicates more extreme CeD disease symptoms. Baseline values was defined as the last observed value before the first dose of gluten.
Time Frame: Baseline and Day 15
Population: The biomarker analysis set consisted of all participants had two endoscopic examinations with biopsies, one before and one after gluten challenge.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group A: Gluten 3 Gram | Group B: Gluten 10 Gram
Number analyzed (Participants) | 7 | 7
ratio
  Baseline | 2.10 (0.697) | 2.30 (0.893)
  Change at Day 15 | -0.06 (0.516) | -1.53 (0.941)
Statistical Analysis 1: Comparison: Group A: Gluten 3 Gram; Gluten 3 gram: Baseline versus Day 15. Change in Vh:Cd follows a normal distribution. A 1-sided paired t-test was used to compare Baseline and follow-up Vh:Cd measures. The normality assumption was checked using the Shapiro-Wilk test. If the data was not normal at alpha=0.05, a 1-sided Wilcoxon signed-rank test was used instead to compare Vh:CdBaseline (B) and Vh:Cd15; Test type: Other; p = 0.385, t-test, 1 sided
Statistical Analysis 2: Comparison: Group B: Gluten 10 Gram; Gluten 10 gram: Baseline versus Day 15. Change in Vh:Cd follows a normal distribution. A 1-sided paired t-test was used to compare Baseline and follow-up Vh:Cd measures. The normality assumption was checked using the Shapiro-Wilk test. If the data was not normal at alpha=0.05, a 1-sided Wilcoxon signed-rank test was used instead to compare Vh:CdB and Vh:Cd15; Test type: Other; p = 0.003, t-test, 1 sided

2. Primary Outcome: Change From Baseline in Small Intestine Histology Based on Intraepithelial Lymphocytes (IEL) Counts
Description: IELs are white blood cells (WBCs) interspersed between epithelial cells of the small and large intestine where they function to preserve the integrity of the mucosal barrier by protecting the epithelium against pathogen or immune-induced pathology. Increased IELs count indicated more extreme CeD disease symptoms. Baseline values was defined as the last observed value before the first dose of gluten.
Time Frame: Baseline and Day 15
Population: The biomarker analysis set consisted of all participants who had two endoscopic examinations with biopsies, one before and one after gluten challenge.
Measure: Mean (Standard Deviation); unit: IEL per 100 epithelial cells
Arm/Group | Group A: Gluten 3 Gram | Group B: Gluten 10 Gram
Number analyzed (Participants) | 7 | 7
IEL per 100 epithelial cells
  Baseline | 26.74 (15.861) | 26.68 (8.248)
  Change at Day 15 | 9.56 (15.206) | 26.80 (14.908)
Statistical Analysis 1: Comparison: Group A: Gluten 3 Gram; Gluten 3 gram: Baseline versus Day 15. The Poisson distribution assumption was checked using Kolmogorov-Smirnov test. Poisson generalized linear mixed models (GLMM) was fitted to data, where IEL measurements were grouped by participant (the random effect) and the change in IEL counts was the fixed effect. If the data was found to not be Poisson at alpha=0.05, a 1-sided Wilcoxon signed-rank test was used instead to compare IELB and IEL15; Test type: Other; p = 0.010, Poisson distribution
Statistical Analysis 2: Comparison: Group B: Gluten 10 Gram; Gluten 10 gram: Baseline versus Day 15. The Poisson distribution assumption was checked using Kolmogorov-Smirnov test. Poisson GLMM was fitted to data, where IEL measurements were grouped by participant (the random effect) and the change in IEL counts was the fixed effect. If the data was found to not be Poisson at alpha=0.05, a 1-sided Wilcoxon signed-rank test was used instead to compare IELB and IEL15; Test type: Other; p = 0.006, Poisson distribution

3. Secondary Outcome: Correlation Coefficient Changes Between Gluten-specific Blood T Cells and Standard CeD Histological Assessments
Description: Standard measures used for diagnosing CeD: Vh:CD ratio and IEL counts. T cell measurements taken before first dose of gluten were correlated with Baseline Vh:Cd ratio and IEL counts, and T cell measurements taken after first dose of gluten were correlated with Day 15 Vh:Cd ratio and IEL counts using Spearman correlation. Villi were small finger like projections that line small intestine, promote nutrient absorption and are often shortened in CeD participants. Crypts were grooves between villi that were often elongated in CeD participants. IELs were WBCs interspersed between epithelial cells of intestine where they function to preserve integrity of mucosal barrier by protecting epithelium against pathogen/immune-induced pathology. Decreased Vh:Cd ratio and increased IELs count indicated more extreme CeD symptoms. Baseline value: last observed value before first dose of gluten. Tr: T cell value taken before first dose of gluten. T6: T cell value at Day 6. T15: T cell value at Day 15.
Time Frame: At Baseline, Days 6 and 15
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Group A: Gluten 3 Gram | Group B: Gluten 10 Gram
Number analyzed (Participants) | 7 | 7
correlation coefficient
  Tr: Baseline Vh:Cd ratio | -0.0355 | 0.1480
  Tr: Baseline IEL counts | -0.0050 | -0.0905
  T6: Day 15 Vh: Cd ratio | 0.0368 | -0.0170
  T6: Day 15 IEL counts | 0.2179 | 0.0595
  T15: Day 15 Vh: Cd ratio | -0.0913 | 0.0214
  T15: Day 15 IEL counts | 0.2967 | 0.0192

4. Secondary Outcome: Change From Baseline in Gluten-specific T Cells in Blood Based on Enzyme-linked Immune Absorbent Spot (ELISPot) Assay and T Cell Receptor (TCR) Human Leukocyte Antigen Serotype (HLA-DQ2)-Tetramers
Description: ELISpot assay and gluten specific TCR measures drug response by quantifying changes in the number or function of gluten-specific T cells. Baseline value was defined as the last observed value before the first dose of gluten.
Time Frame: Baseline and Day 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: per million CD4+ T cells
Arm/Group | Group A: Gluten 3 Gram | Group B: Gluten 10 Gram
Number analyzed (Participants) | 7 | 7
per million CD4+ T cells
  Baseline (ELISpot) | 1.00 (1.956) | 1.45 (1.756)
  Change at Day 6 (ELISpot) | 3.83 (6.902) | 25.12 (29.025)
  Baseline (Tetramer) | 34.62 (29.215) | 17.33 (14.894)
  Change at Day 6 (Tetramer) | 26.76 (54.084) | 522.47 (788.177)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) are adverse events that started after the first dose of gluten up to Day 43
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Group A: Gluten 3 Gram | Group B: Gluten 10 Gram
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 3/9 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Gluten 3 Gram (N=9) | Group B: Gluten 10 Gram (N=7)
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gluten sensitivity (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT03409796/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT03409796/SAP_001.pdf